CLINICAL TRIAL: NCT01576744
Title: Serum Concentration of HE4, a New Marker for Ovarian Cancer, Changes Little Throughout IVF Stimulation
Brief Title: Serum Biomarker HE4 During IVF Treatment
Acronym: FHE4
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Antti Perheentupa, Associate Professor, Turku University Hospital
Other Study IDs: FHE4-2010
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-06

CONDITIONS: IVF Treatment; Human Epididymal Secretory Protein E4
Keywords: HE4; IVF; Biomarker; Ovarian cancer; Infertility
MeSH Terms: conditions — Ovarian Neoplasms; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Repeated serum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Human epididymal secretory protein 4 (HE4) is a new biomarker for ovarian cancer. The effect of IVF stimulation will be evaluated in order to see whether severe hormonal changes in the gonadotrophin and steroid status affect the serum levels of this marker. Findings will be compared to serum concentrations of CA-125, which is currently the most often used marker for ovarian cancer.

The intention is to determine the serum concentration of HE4 and CA-125 in serial samples in 20 women undergoing IVF stimulation. Samples will be taken following GnRH agonist suppression, 2-3 times during FSH stimulation, at ovum pick up and two weeks following embryo transfer at the time of the hCG-test. The ovarian follicle count and the serum estradiol concentrations are recorded throughout the treatment. The serum biomarker HE4 is expected to ba a stable marker, which does not respond significantly to hormonal stimulation.

ELIGIBILITY:
Inclusion Criteria:

* infertility treated by IVF

Exclusion Criteria:

* pelvic tumor
* overweight (BMI over 35)

Ages: 27 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Finnish caucasian women being treated for infertility by in vitro-fertilization
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Antti H Perheentupa, MD, PhD, Principal Investigator — Department of Obstetrics and Gynecology, Turku University Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Turku University Hospital, Turku, Finland